CLINICAL TRIAL: NCT06390254
Title: Effectiveness of a Resilience-Building Nursing Intervention on Psychological Well-being in Community-Dwelling Older Adults
Brief Title: Resilience-Building Nursing Intervention for Elderly Well-being
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Shaban, Clinical Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RBNI-PWB-001
Record Dates: First submitted 2024-04-21; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Psychological Well-being in Older Adults; Resilience Building Intervention; Community Dwelling Older Adults
Keywords: Resilience; Psychological well-being; Older adults; Nursing intervention; Community-dwelling; Geriatrics; Quality of life
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The interventional study model for this trial follows a randomized controlled design. Participants will be randomly assigned to either the intervention group or the control group. The intervention group will receive the resilience-building nursing intervention, while the control group will receive standard care. This design allows for a rigorous evaluation of the effectiveness of the intervention by comparing outcomes between the two groups. Blinding of participants and investigators may or may not be feasible depending on the nature of the intervention. The study will adhere to established protocols for randomization, allocation concealment, and blinding to minimize bias and ensure the validity of the findings.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- resilience-building nursing intervention. (Experimental): Participants receiving the resilience-building nursing intervention.
  Interventions: Other: Resilience-Enhancing Nursing Suppor
- Control (No Intervention): Participants receiving standard care or placebo, depending on the design of your study.

INTERVENTIONS:
Other: Resilience-Enhancing Nursing Suppor — The resilience-building nursing intervention in this study is a multifaceted approach aimed at enhancing the psychological well-being and coping abilities of community-dwelling older adults. Unlike standard care, which typically focuses on symptom management, this intervention emphasizes proactive strategies to promote resilience and improve overall quality of life.
  Arms: resilience-building nursing intervention.

SUMMARY:
The objective of this study is to evaluate the impact of a resilience-enhancing nursing intervention on the psychological well-being of older adults living in the community. Participants will benefit from individualized nursing support designed to bolster their resilience and coping skills. This intervention will be customized to meet personal requirements and provided in a nurturing setting. Engaging in this study could result in enhanced well-being and life quality. Although some minor discomforts may arise during assessments or interventions, the confidentiality and rights of the participants will be rigorously safeguarded.

DETAILED DESCRIPTION:
Background:

As the global population ages, there is an increasing need to address the psychological well-being of older adults living independently in the community. Previous research has highlighted the importance of resilience in maintaining mental health and coping with life stressors among older individuals. However, there is limited evidence on the effectiveness of specific interventions aimed at enhancing resilience in this population.

Objective:

The primary objective of this study is to evaluate the effectiveness of a resilience-building nursing intervention in improving the psychological well-being of community-dwelling older adults. Secondary objectives include assessing the impact of the intervention on factors such as social support, coping strategies, and quality of life.

Study Design:

This study will employ a randomized controlled trial design. Participants will be randomly assigned to either the intervention group, receiving the resilience-building nursing intervention, or the control group, receiving standard care.

Intervention:

The resilience-building nursing intervention will consist of individualized sessions delivered by trained nurses. The intervention will focus on enhancing participants' resilience through skill-building exercises, cognitive-behavioral techniques, and psychoeducation. Sessions will be tailored to address the unique needs and challenges of each participant.

Participants:

The target population for this study includes community-dwelling older adults aged 65 and above who are experiencing mild to moderate psychological distress. Participants will be recruited from community centers, senior living facilities, and primary care clinics.

Procedures:

Participants will undergo baseline assessments to collect demographic information and baseline measures of psychological well-being. Those assigned to the intervention group will receive the resilience-building nursing intervention over a specified period, with follow-up assessments conducted at regular intervals to evaluate outcomes.

Outcome Measures:

Primary outcome measures will include changes in psychological well-being, as assessed by standardized scales such as the Geriatric Depression Scale and the Psychological Well-being Scale. Secondary outcome measures will include social support, coping strategies, and quality of life.

Statistical Analysis:

Data will be analyzed using appropriate statistical methods, including t-tests, chi-square tests, and linear regression. Sample size calculations will ensure adequate power to detect meaningful differences between groups.

Ethical Considerations:

This study will adhere to ethical principles outlined in the Declaration of Helsinki. Informed consent will be obtained from all participants, and measures will be taken to ensure participant confidentiality and privacy.

Data Management:

Data will be collected using secure electronic data capture systems and stored in accordance with institutional guidelines and data protection regulations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 60 years and older.
* Individuals living in the community.
* Mild to moderate psychological distress.

Exclusion Criteria:

* Severe cognitive impairment or dementia.
* Significant medical or psychiatric comorbidities that could impede participation in the intervention.
* Inability to understand and communicate in the language used for the intervention materials.
* Concurrent participation in another research study involving psychological interventions.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-25 (Estimated); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Psychological Well-being Assessment | Psychological well-being will be assessed at baseline, prior to the intervention, and at follow-up assessments conducted at 1 months post-intervention.
  The main outcome measure of this study is the alteration in psychological well-being among participants, gauged using standardized the Psychological Well-being Scale (PWB)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zahid N, Martins RS, Zahid W, Khalid W, Azam I, Bhamani SS, Ahmad K, Jabbar A, Shamim MS, Khan RJ, Javed G, Bari E, Asad N, Enam SA. Resilience and its associated factors in brain tumor patients in Karachi, Pakistan: An analytical cross-sectional study. Psychooncology. 2021 Jun;30(6):882-891. doi: 10.1002/pon.5661. Epub 2021 Mar 10. PMID 33609048
- [Result] Wu Y, Dai Z, Jing S, Liu X, Zhang L, Liu X, Ren T, Fu J, Chen X, Xiao W, Wang H, Huang Y, Wang W, Gu X, Ma L, Zhang S, Yu Y, Li L, Han Z, Su X, Qiao Y. Prevalence and influencing factors of PTSD symptoms among healthcare workers: A multicenter cross-sectional study during the surge period of the COVID-19 pandemic since December 2022 in the Chinese mainland. J Affect Disord. 2024 Mar 1;348:70-77. doi: 10.1016/j.jad.2023.12.008. Epub 2023 Dec 6. PMID 38065482
- [Result] Jayakrishnan K, Baruah A, Kumar P, Javeth A. Scales and Interventions for Resilience among Treatment-Seeking Patients with Depression: A Systematic Review. J Caring Sci. 2023 May 21;12(2):84-93. doi: 10.34172/jcs.2023.31964. eCollection 2023 Jun. PMID 37469753
- [Result] Cleary M, Kornhaber R, Thapa DK, West S, Visentin D. The effectiveness of interventions to improve resilience among health professionals: A systematic review. Nurse Educ Today. 2018 Dec;71:247-263. doi: 10.1016/j.nedt.2018.10.002. Epub 2018 Oct 11. PMID 30342300
- [Result] Chow KM, Tang FWK, Tang WPY, Leung AWY. Resilience-building module for undergraduate nursing students: A mixed-methods evaluation. Nurse Educ Pract. 2020 Nov;49:102912. doi: 10.1016/j.nepr.2020.102912. Epub 2020 Nov 6. PMID 33186821
- [Result] Henshall C, Davey Z, Srikesavan C, Hart L, Butcher D, Cipriani A. Implementation of a Web-Based Resilience Enhancement Training for Nurses: Pilot Randomized Controlled Trial. J Med Internet Res. 2023 Feb 14;25:e43771. doi: 10.2196/43771. PMID 36787181